CLINICAL TRIAL: NCT04365725
Title: Multicenter, Retrospective Study of the Effects of Remdesivir in the Treatment of Severe Covid-19 Infections.
Acronym: REMDECO-19
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200522
Record Dates: First submitted 2020-04-25; First posted 2020-04-28 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: COVID-19
Keywords: COVID-19; Remdesivir
MeSH Terms: conditions — COVID-19 | interventions — remdesivir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Remdesivir — Compassionate provision

SUMMARY:
This study is a retrospective cohort trial to assess the efficacy of remdesivir in hospitalized adult patients diagnosed with COVID-19. The study is a multicenter trial which will be carried out on different sites in France. This trial is retrospective and will analyze the data collected during treatment.

DETAILED DESCRIPTION:
COVID-19 is a respiratory disease caused by a new coronavirus (SARS-CoV-2) and causes significant morbidity and mortality. There is currently no approved treatment for the treatment of patients with COVID-19. Global efforts to evaluate new antivirals and therapeutic strategies to treat COVID-19 have intensified. To quickly propose a first line of defense and fight against the virus in hospitalized patients, the World Health Organization (WHO) relies on already existing drugs, "repositioned", which are immediately available in large quantities and present a good security profile. Remdesivir (GS-5734) is a broad spectrum nucleotide analogue that inhibits RNA-dependent RNA polymerase activity among a diverse group of RNA viruses. Non-clinical and clinical data suggest that remdesivir may be useful for the treatment of COVID-19. WHO has identified remdesivir as a candidate drug of interest to be studied in clinical trials. Compassionate provision of the drug allowed its use before clinical trials began. This retrospective cohort study is designed to analyze the data collected during the routine care of patients who have benefited from this compassionate provision.

The data collected in real life during care will allow a multivariate analysis quickly providing elements of response on a typology of patients and level of progression of the disease for which remdesivir would bring a more or less significant clinical benefit. Multivariate analysis of these data will allow the identification of variables at the initiation of treatment with remdesivir that are potentially predictive of its clinical efficacy.

The period for collecting data collected during treatment for an individual subject is 30 days. The retrospective collection begins on the day before initiation of treatment with remdesivir up to 29 days after. A note of information and of no objection to the collection of data will be sent to the patient. The data collected comes from the patient's medical records. The observations will be entered by investigative doctors and or clinical study technicians.

Statistical analysis will be carried out using SAS 9.3 and / or R software. All the analyzes carried out will follow the recommendations of STROBE for observational studies. A detailed statistical analysis plan will be carried out before basic freezing and data analysis. Quantitative data will be described as the mean and standard deviation or medians and quartiles depending on the distribution of the data. Qualitative data will be described in terms of numbers and percentages. Comparisons of quantitative data will be analyzed using the student or wilcoxon test depending on the test application conditions, and comparisons of categorical variables will be made using the Chi2 or Fisher test, if appropriate. Multivariate models will be produced to explore the factors associated with patient prognosis. The clinical development of patients described on a 7-point ordinal scale will be divided into two in order to create logistic models. The entire process of selecting variables in the models will be described in the analysis plan which will be validated before the database freezes.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years old.
* SARS-CoV-2 infection confirmed.
* Hospitalized patients who received at least one administration of remdesivir therapy outside of clinical trials

Exclusion Criteria:

* Patients included in a clinical trial testing remdesivir as an investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult hospital patients diagnosed with COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Clinical course on Day 15. | 15 days
  Study the prognostic factors of the clinical course of patients on Day 15 under treatment with remdesivir. Clinical progress will be categorized using a 7-point ordinal scale.

SECONDARY OUTCOMES:
Clinical course on Day 3. | 3 days
  Explore the prognostic factors of the clinical course of patients on Day 3
Clinical course on Day 8 | 8 days
  Explore the prognostic factors of the clinical course of patients on Day 8
Clinical course on Day 11. | 11 days
  Explore the prognostic factors of the clinical course of patients on Day11
Clinical course on Day 29. | 29 days
  Explore the prognostic factors of the clinical course of patients on D29.
Duration of treatment | 29 days
  Duration of treatment with remdesivir
Sepsis-related Organ Failure Assessment score | Day 3, 8, 11, 15 and 29
  PaO2 / FiO2 and artificial ventilation; platelets; bilirubin; average blood pressure and use of vasoactive drugs; Glasgow score; creatinine.
Duration without mechanical ventilation | 29 days
  Duration without mechanical ventilation within 29 days of initiation of treatment with remdesivir
Mortality | 29 days
  Mortality at 29 days after initiation of treatment with remdesivir.
cumulative incidence of grade 3 and 4 adverse events (AEs). | 29 days
  Evaluate the safety of the treatment with cumulative incidence of grade 3 and 4 adverse events (AEs).

CONTACTS AND LOCATIONS:
Overall Officials: Jérémie ZERBIT, PharmaD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Chan JF, Kok KH, Zhu Z, Chu H, To KK, Yuan S, Yuen KY. Genomic characterization of the 2019 novel human-pathogenic coronavirus isolated from a patient with atypical pneumonia after visiting Wuhan. Emerg Microbes Infect. 2020 Jan 28;9(1):221-236. doi: 10.1080/22221751.2020.1719902. eCollection 2020. PMID 31987001
- [Background] Wu JT, Leung K, Leung GM. Nowcasting and forecasting the potential domestic and international spread of the 2019-nCoV outbreak originating in Wuhan, China: a modelling study. Lancet. 2020 Feb 29;395(10225):689-697. doi: 10.1016/S0140-6736(20)30260-9. Epub 2020 Jan 31. PMID 32014114
- [Background] Friberg LE, Guedj J. Acute bacterial or viral infection-What's the difference? A perspective from PKPD modellers. Clin Microbiol Infect. 2020 Sep;26(9):1133-1136. doi: 10.1016/j.cmi.2019.12.008. Epub 2019 Dec 31. No abstract available. PMID 31899337
- [Background] Goncalves A, Bertrand J, Ke R, Comets E, de Lamballerie X, Malvy D, Pizzorno A, Terrier O, Rosa Calatrava M, Mentre F, Smith P, Perelson AS, Guedj J. Timing of Antiviral Treatment Initiation is Critical to Reduce SARS-CoV-2 Viral Load. CPT Pharmacometrics Syst Pharmacol. 2020 Sep;9(9):509-514. doi: 10.1002/psp4.12543. Epub 2020 Aug 7. PMID 32558354
- [Background] Lo MK, Jordan R, Arvey A, Sudhamsu J, Shrivastava-Ranjan P, Hotard AL, Flint M, McMullan LK, Siegel D, Clarke MO, Mackman RL, Hui HC, Perron M, Ray AS, Cihlar T, Nichol ST, Spiropoulou CF. GS-5734 and its parent nucleoside analog inhibit Filo-, Pneumo-, and Paramyxoviruses. Sci Rep. 2017 Mar 6;7:43395. doi: 10.1038/srep43395. PMID 28262699
- [Background] Lo MK, Feldmann F, Gary JM, Jordan R, Bannister R, Cronin J, Patel NR, Klena JD, Nichol ST, Cihlar T, Zaki SR, Feldmann H, Spiropoulou CF, de Wit E. Remdesivir (GS-5734) protects African green monkeys from Nipah virus challenge. Sci Transl Med. 2019 May 29;11(494):eaau9242. doi: 10.1126/scitranslmed.aau9242. PMID 31142680
- [Background] Warren TK, Jordan R, Lo MK, Ray AS, Mackman RL, Soloveva V, Siegel D, Perron M, Bannister R, Hui HC, Larson N, Strickley R, Wells J, Stuthman KS, Van Tongeren SA, Garza NL, Donnelly G, Shurtleff AC, Retterer CJ, Gharaibeh D, Zamani R, Kenny T, Eaton BP, Grimes E, Welch LS, Gomba L, Wilhelmsen CL, Nichols DK, Nuss JE, Nagle ER, Kugelman JR, Palacios G, Doerffler E, Neville S, Carra E, Clarke MO, Zhang L, Lew W, Ross B, Wang Q, Chun K, Wolfe L, Babusis D, Park Y, Stray KM, Trancheva I, Feng JY, Barauskas O, Xu Y, Wong P, Braun MR, Flint M, McMullan LK, Chen SS, Fearns R, Swaminathan S, Mayers DL, Spiropoulou CF, Lee WA, Nichol ST, Cihlar T, Bavari S. Therapeutic efficacy of the small molecule GS-5734 against Ebola virus in rhesus monkeys. Nature. 2016 Mar 17;531(7594):381-5. doi: 10.1038/nature17180. Epub 2016 Mar 2. PMID 26934220
- [Background] Mulangu S, Dodd LE, Davey RT Jr, Tshiani Mbaya O, Proschan M, Mukadi D, Lusakibanza Manzo M, Nzolo D, Tshomba Oloma A, Ibanda A, Ali R, Coulibaly S, Levine AC, Grais R, Diaz J, Lane HC, Muyembe-Tamfum JJ; PALM Writing Group; Sivahera B, Camara M, Kojan R, Walker R, Dighero-Kemp B, Cao H, Mukumbayi P, Mbala-Kingebeni P, Ahuka S, Albert S, Bonnett T, Crozier I, Duvenhage M, Proffitt C, Teitelbaum M, Moench T, Aboulhab J, Barrett K, Cahill K, Cone K, Eckes R, Hensley L, Herpin B, Higgs E, Ledgerwood J, Pierson J, Smolskis M, Sow Y, Tierney J, Sivapalasingam S, Holman W, Gettinger N, Vallee D, Nordwall J; PALM Consortium Study Team. A Randomized, Controlled Trial of Ebola Virus Disease Therapeutics. N Engl J Med. 2019 Dec 12;381(24):2293-2303. doi: 10.1056/NEJMoa1910993. Epub 2019 Nov 27. PMID 31774950
- [Background] Sheahan TP, Sims AC, Graham RL, Menachery VD, Gralinski LE, Case JB, Leist SR, Pyrc K, Feng JY, Trantcheva I, Bannister R, Park Y, Babusis D, Clarke MO, Mackman RL, Spahn JE, Palmiotti CA, Siegel D, Ray AS, Cihlar T, Jordan R, Denison MR, Baric RS. Broad-spectrum antiviral GS-5734 inhibits both epidemic and zoonotic coronaviruses. Sci Transl Med. 2017 Jun 28;9(396):eaal3653. doi: 10.1126/scitranslmed.aal3653. PMID 28659436
- [Background] Sheahan TP, Sims AC, Leist SR, Schafer A, Won J, Brown AJ, Montgomery SA, Hogg A, Babusis D, Clarke MO, Spahn JE, Bauer L, Sellers S, Porter D, Feng JY, Cihlar T, Jordan R, Denison MR, Baric RS. Comparative therapeutic efficacy of remdesivir and combination lopinavir, ritonavir, and interferon beta against MERS-CoV. Nat Commun. 2020 Jan 10;11(1):222. doi: 10.1038/s41467-019-13940-6. PMID 31924756
- [Background] Agostini ML, Andres EL, Sims AC, Graham RL, Sheahan TP, Lu X, Smith EC, Case JB, Feng JY, Jordan R, Ray AS, Cihlar T, Siegel D, Mackman RL, Clarke MO, Baric RS, Denison MR. Coronavirus Susceptibility to the Antiviral Remdesivir (GS-5734) Is Mediated by the Viral Polymerase and the Proofreading Exoribonuclease. mBio. 2018 Mar 6;9(2):e00221-18. doi: 10.1128/mBio.00221-18. PMID 29511076
- [Background] de Wit E, Rasmussen AL, Falzarano D, Bushmaker T, Feldmann F, Brining DL, Fischer ER, Martellaro C, Okumura A, Chang J, Scott D, Benecke AG, Katze MG, Feldmann H, Munster VJ. Middle East respiratory syndrome coronavirus (MERS-CoV) causes transient lower respiratory tract infection in rhesus macaques. Proc Natl Acad Sci U S A. 2013 Oct 8;110(41):16598-603. doi: 10.1073/pnas.1310744110. Epub 2013 Sep 23. PMID 24062443
- [Background] de Wit E, Feldmann F, Cronin J, Jordan R, Okumura A, Thomas T, Scott D, Cihlar T, Feldmann H. Prophylactic and therapeutic remdesivir (GS-5734) treatment in the rhesus macaque model of MERS-CoV infection. Proc Natl Acad Sci U S A. 2020 Mar 24;117(12):6771-6776. doi: 10.1073/pnas.1922083117. Epub 2020 Feb 13. PMID 32054787
- [Background] Wang M, Cao R, Zhang L, Yang X, Liu J, Xu M, Shi Z, Hu Z, Zhong W, Xiao G. Remdesivir and chloroquine effectively inhibit the recently emerged novel coronavirus (2019-nCoV) in vitro. Cell Res. 2020 Mar;30(3):269-271. doi: 10.1038/s41422-020-0282-0. Epub 2020 Feb 4. No abstract available. PMID 32020029
- [Background] Grein J, Ohmagari N, Shin D, Diaz G, Asperges E, Castagna A, Feldt T, Green G, Green ML, Lescure FX, Nicastri E, Oda R, Yo K, Quiros-Roldan E, Studemeister A, Redinski J, Ahmed S, Bernett J, Chelliah D, Chen D, Chihara S, Cohen SH, Cunningham J, D'Arminio Monforte A, Ismail S, Kato H, Lapadula G, L'Her E, Maeno T, Majumder S, Massari M, Mora-Rillo M, Mutoh Y, Nguyen D, Verweij E, Zoufaly A, Osinusi AO, DeZure A, Zhao Y, Zhong L, Chokkalingam A, Elboudwarej E, Telep L, Timbs L, Henne I, Sellers S, Cao H, Tan SK, Winterbourne L, Desai P, Mera R, Gaggar A, Myers RP, Brainard DM, Childs R, Flanigan T. Compassionate Use of Remdesivir for Patients with Severe Covid-19. N Engl J Med. 2020 Jun 11;382(24):2327-2336. doi: 10.1056/NEJMoa2007016. Epub 2020 Apr 10. PMID 32275812
- [Background] Chan JF, Yuan S, Kok KH, To KK, Chu H, Yang J, Xing F, Liu J, Yip CC, Poon RW, Tsoi HW, Lo SK, Chan KH, Poon VK, Chan WM, Ip JD, Cai JP, Cheng VC, Chen H, Hui CK, Yuen KY. A familial cluster of pneumonia associated with the 2019 novel coronavirus indicating person-to-person transmission: a study of a family cluster. Lancet. 2020 Feb 15;395(10223):514-523. doi: 10.1016/S0140-6736(20)30154-9. Epub 2020 Jan 24. PMID 31986261
- [Result] Beigel JH, Tomashek KM, Dodd LE, Mehta AK, Zingman BS, Kalil AC, Hohmann E, Chu HY, Luetkemeyer A, Kline S, Lopez de Castilla D, Finberg RW, Dierberg K, Tapson V, Hsieh L, Patterson TF, Paredes R, Sweeney DA, Short WR, Touloumi G, Lye DC, Ohmagari N, Oh MD, Ruiz-Palacios GM, Benfield T, Fatkenheuer G, Kortepeter MG, Atmar RL, Creech CB, Lundgren J, Babiker AG, Pett S, Neaton JD, Burgess TH, Bonnett T, Green M, Makowski M, Osinusi A, Nayak S, Lane HC; ACTT-1 Study Group Members. Remdesivir for the Treatment of Covid-19 - Final Report. N Engl J Med. 2020 Nov 5;383(19):1813-1826. doi: 10.1056/NEJMoa2007764. Epub 2020 Oct 8. PMID 32445440